CLINICAL TRIAL: NCT01847456
Title: Influence of Brain Insulin Sensitivity on Peripheral Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, andreas fritsche, Professor of Medicine, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SFB 997 A01 WP7
Record Dates: First submitted 2013-04-28; First posted 2013-05-06 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Insulin Sensitivity
Keywords: whole body insulin sensitivity; insulin action in the brain
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- insulin nasal spray (Experimental): 160 Units of human insulin as nasal spray
  Interventions: Drug: human insulin as nasal spray
- Placebo nasal spray (Placebo Comparator): Nasalspray containing placebo solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: human insulin as nasal spray
  Arms: insulin nasal spray
Drug: Placebo
  Arms: Placebo nasal spray

SUMMARY:
The researchers will investigate if brain insulin action influences peripheral insulin sensitivity in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 28 kg/m2
* normal HbA1c
* healthy volunteers

Exclusion Criteria:

* Heparin induced thrombocytopenia (HIT)
* metal implants
* cardial diseases
* anemia
* patients taking any kind of drugs

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity as measured by clamp | 45 minutes to 120 minutes post nasal spray
  We will measure insulin sensitivity by hyperinsulinemic euglycemic clamp before and after nasal spray application. We will compare the post-spray insulin sensitivity between the two condition (insulin nasal spray vs placebo nasal spray). Furthermore, we will compare insulin sensitivity before and after nasal insulin application.

SECONDARY OUTCOMES:
Autonomous nervous system activity | 45 to 120 minutes post spray
  Activity of the autonomous nervous system will be estimated by heart rate variability in ECG. We will compare the post-spray autonomous nervous system activity between the two condition (insulin nasal spray vs placebo nasal spray). Furthermore, we will compare autonomous nervous system activity before and after nasal insulin application.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Internal medicine IV, Tübingen, Germany

REFERENCES:
- [Derived] Heni M, Wagner R, Kullmann S, Veit R, Mat Husin H, Linder K, Benkendorff C, Peter A, Stefan N, Haring HU, Preissl H, Fritsche A. Central insulin administration improves whole-body insulin sensitivity via hypothalamus and parasympathetic outputs in men. Diabetes. 2014 Dec;63(12):4083-8. doi: 10.2337/db14-0477. Epub 2014 Jul 15. PMID 25028522